CLINICAL TRIAL: NCT01622114
Title: Evaluation of the Association Between the Menstrual Cycle and Weight Loss in Healthy, Overweight Premenopausal Women - A 6-Month Intervention
Brief Title: Evaluation of the Association Between the Menstrual Cycle and Weight Loss in Healthy, Overweight Premenopausal Women
Acronym: MENSTRALEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, Dr Med, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: B252
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: Obesity; Weight reduction; premenopausal Women; Menstrual cycle; quality of life; food cravings
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menstralean group (Experimental): Represents a program which is designed to induce weight loss by taking into account the physiology of each menstrual phase in terms of adjusting diet and physical activity to the body's cyclic changes in energy demands.
  The diet will be adjusted to match one menstrual cycle in duration (approx. 1 month) and will be separated into three phases corresponding to three menstrual phases: menstruation (days 1-5), the follicular phase (days 6-14), and the luteal phase (days 15-28). All women in this group will start the program at day 1 in their cycle. The diet will be repeated six times for each woman, which equals six months.
  Interventions: Other: Evaluation of the Association between the Menstrual Cycle and Weight Loss in Healthy, Overweight Premenopausal Women
- Control Group: (Active Comparator): Represents a program where subjects engage in a similar diet and exercise program as the Menstralean Group, specifically based on the educational diet system "Eat for Life". Importantly, the subjects in Control group will start the program at a random time in their menstrual cycles.
  Eat for Life is a simple tool for controlling the energy content and nutritional composition of your diet. The method is based on a system of counters that ensure strict control of the diet whilst still allowing a great deal of freedom of choice. The subjects in the Control Group will also receive exactly the same attention and undergo the same visits and measurements as the Menstralean Group.
  Interventions: Other: Evaluation of the Association between the Menstrual Cycle and Weight Loss in Healthy, Overweight Premenopausal Women

INTERVENTIONS:
Other: Evaluation of the Association between the Menstrual Cycle and Weight Loss in Healthy, Overweight Premenopausal Women — 2-arm parallel 6 month study with the obejective to examine the impact of the menstrual cycle on weight loss attempts in healthy overweight premenopausal women randomized to two different weight management programs. The women may not use hormonal contraceptive agents other than an IUD.

SUMMARY:
Achievement and maintenance of weight loss in obese individuals has proven difficult. Many hypotheses have suggested potential biological mechanisms to explain why weight loss attempts often fail, and the surrounding obesogenic environment also seems an obvious candidate. Among the biological factors proposed is gender, and weight loss trials have frequently shown that females are less successful than males at losing weight and at maintaining weight loss.

Women's weight is influenced by the menstrual cycle, in which changes in hormonal levels and interactions work to modulate fertility. These hormones control the menstrual cycle and coordinate the required changes in energy intake, expenditure, and storage, whilst preparing the body for pregnancy every month. As reproduction is a primary biological function, these hormones may be such strong mediators of eating behavior that they influence the outcome of a weight loss attempt. The menstrual cycle should therefore be taken into consideration as a factor in the physiology of energy balance in premenopausal women.

The cycle can be divided into three phases: menstruation or early follicular phase (days 1-5), late follicular phase that lasts until ovulation (~days 6-14, and the luteal phase (days 15-28).

Studies have shown that in the luteal phase of the menstrual cycle, women's energy intake and energy expenditure are increased and women experience more frequent cravings for foods, particularly those high in carbohydrate and fat, than during the follicular phase. A trend towards reduced carbohydrate utilization and increased fat oxidation in the luteal phase has also been reported, together with prolonged time to exhaustion when exercising at submaximal intensities. This suggests that the potential of the underlying physiology related to each phase of the menstrual cycle may be worth considering as an element in strategies to optimize weight loss.

In 2010 the investigators carried out a 90-day randomized, controlled pilot study in order to gain feedback on and assess acceptance of the meal and exercise plans being used and to observe if less control visits than planed in the main study were sufficient to achieve good compliance. Twenty eight were sreened and 24 were included. Subjects were randomized to either program A (given meal and exercise plans in relation to phases of their menstrual cycles) or Program B (a reduced calorie diet, calorie-matched to program A). The pilot study showed that Group A (The Menstralean group) tended to have a greater average weight loss at 60 days (-5.29 vs -3.57 kg, p = 0.06) and 90 days (-4.22 vs -2.75 kgs, p = 0.2) compared to the control groups. There was a dropout rate of 27%. This was primarily due to an inadequate number of control visits and contact with the subjects. Thus the Menstralean program seems to have the potential to enhance weight loss in overweight and obese women. However, the main study has to be carried out with more subjects in each group in a longer duration and with more support and contact with the subjects.

The aim of the present trial is to examine the impact of the menstrual cycle on weight loss attempts in healthy overweight (BMI > 27 kg/m2) premenopausal women (18-40 years) randomized to two different weight management programs for a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females between the ages of 18-40 (inclusive)
* BMI > 27 kg/m².
* Regular menstrual cycle (28 ± 4 days - with a maximum of 4 days within-subject variation in menstrual cycle duration.
* Weight stable (within ± 3-kg) 2 months prior to study inclusion
* Must use barrier contraception (e.g. male/female condom) for the study's duration
* Must be willing to follow the prescribed diet/exercise plan for the study's duration

Exclusion Criteria:

* On hormonal contraceptives (IUD are allowed) or any other daily use of medications which can make the subject unsuitable for inclusion in the study.
* Any significant health problem (history of cancer, HIV/AIDS, Diabetes, cardiovascular disease, untreated hypothyroidism, etc.)
* Restrictions against participating in cardiovascular exercise and strength training
* Any condition, which in the opinion of the investigator makes the subject unsuitable for inclusion in the study.
* Women who are pregnant,lactating, or planning to become pregnant during the study period

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in body weight (kg) | will be measured at baseline and week 2, 4, 8, 12, 16, 20, 24 and at follow up (8 months after initiation)
  Assessment of body weight will be carried on a digital scale to the nearest 0.05 kg. The measurement will be carried out after the subjects have emptied their bladder and only wearing underwear.

SECONDARY OUTCOMES:
Change in waist circumference (cm) | measurement will be carried out at baseline and week 2, 12, 24 and at follow up (8 months after initiation)
  Assessment of waist circumference will be carried with a measuring tape to the nearest 0.5 cm. The measurement will be carried out after the subjects have emptied their bladder and only wearing underwear.
Height (cm) | measurement will be carried out at screening
  Height of the subject will measured in a up-right position without shoes to the nearest 0.5 cm.
Change in body mass index (BMI) | measurement will be carried out at baseline and week 2, 4, 8, 12, 16, 20, 24 and at follow up (8 months after initiation)
  BMI is based on the measurement of height and body weight: weight (kg)/ (height (cm)* height (cm))
Assessment of Well-being/quality of life | measurement will be carried out at screening, baseline and week 12 and 24 and after 8 months (follow up)
  Quality of life will be assessed by IWQOL-Lite questionnaire at screening, baseline, week 12, week 24 and at follow-up 8 month after initiation of intervention.
Assessment of Impact of Weight on Quality of Life | measurement will be carried out at screening, baseline and week 12 and 24 and after 8 months (follow up)
  'Impact of Weight on Quality of Life' will be assessed by IWQOL-Lite questionnaire at screening, baseline, week 12, week 24 and at follow-up 8 month after initiation of intervention.
Assessment of Food cravings | measurement will be carried out at screening, baseline and week 12 and 24 and after 8 months (follow up)
  'Impact of Weight on Quality of Life' will be assessed by FCI-II questionnaire at screening, baseline, week 12, week 24 and at follow-up 8 month after initiation of intervention.
Drop-out rate during the first 24 weeks | measured during the 24-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Dr Med, Principal Investigator — Department of Human Nutrition, Faculty of Science, University of Copenhagen, Denmark
Locations (1):
- Department of Human Nutrition, Faculty of Science, University of Copenhagen, Denmark, Frederiksberg, Denmark

REFERENCES:
- [Derived] Geiker NR, Ritz C, Pedersen SD, Larsen TM, Hill JO, Astrup A. A weight-loss program adapted to the menstrual cycle increases weight loss in healthy, overweight, premenopausal women: a 6-mo randomized controlled trial. Am J Clin Nutr. 2016 Jul;104(1):15-20. doi: 10.3945/ajcn.115.126565. Epub 2016 Jun 8. PMID 27281304